CLINICAL TRIAL: NCT02125396
Title: Adjuvant Radiotherapy Comparing Transarterial Chemoembolization for Curative Hepatocellular Carcinoma: a Randomized Controlled Trials
Brief Title: Adjuvant Radiotherapy Comparing TACE for Curative HCC
Acronym: ARTC-HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Affiliated Tumor Hospital, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTC-HCC
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; liver cancer; transarterial chemoembolization; radiotherapy; adjuvant therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Experimental): Adjuvant radiotherapy is used for postoperative curative HCC
  Interventions: Other: Transarterial chemoembolization; Other: Radiotherapy
- Transarterial chemoembolization (Active Comparator): Adjuvant transarterial chemoembolization [5-15 ml lipiodol 5-fluorouracil (500 mg/m2) and adriamycin (30 mg/m2)]
  Interventions: Other: Transarterial chemoembolization; Other: Radiotherapy

INTERVENTIONS:
Other: Transarterial chemoembolization — Adjuvant transarterial chemoembolization [5-15 ml lipiodol 5-fluorouracil (500 mg/m2) and adriamycin (30 mg/m2)]
Other: Radiotherapy — Adjuvant radiotherapy is used for postoperative curative HCC

SUMMARY:
Despite advances in our understanding of hepatocellular carcinoma (HCC) and its diagnosis, the prognosis for patients with HCC remains disheartening, due to a high recurrence rate and frequent intrahepatic metastasis. Various therapies for use after hepatic resection have been reported, but they are associated with adverse side effects or they fail to improve overall survival. Nowadays, adjuvant transarterial chemoembolization (TACE) is recommended as the most effective therapy for postoperative HCC. And the indication is patients with risk factors of recurrence. While more and more prospective studies revealed that radiotherapy is effective for advanced HCC. And the side effects of radiotherapy are controlled. Until now, no prospective or retrospective study compared the efficacy of adjuvant TACE and radiotherapy for postoperative HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Diagnosis of HCC was confirmed by histopathological examination of surgical samples in all patients
* Patients have Child-Pugh A liver function and undergo potentially curative hepatic resection
* Patients with risk factors for recurrence (tumor size >5 cm, multiple nodules, vascular invasion, absence of tumor capsule, poorly differentiated tumor, and narrow resection margin)
* No previous treatment of HCC except liver resection
* No evidence of metastasis to the lymph nodes and/or distant metastases on the basis of preoperative imaging results and perioperative findings
* No malignancy other than HCC for 5 years prior to the initial HCC treatment
* No imaging evidence of invasion into the major portal/hepatic vein branches
* No history of encephalopathy, ascites refractory to diuretics or variceal bleeding

Exclusion Criteria:

* History of cardiac disease:

  * congestive heart failure > New York Heart Association (NYHA) class 2;
  * active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted);
  * cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers, calcium channel blocker or digoxin; or
  * uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of 3 antihypertensive drugs).
* Active clinically serious infections ( > grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
* Excluded therapies and medications, previous and concomitant:

  * Prior use of any systemic anti-cancer treatment for HCC, eg. chemotherapy, immunotherapy or hormonal therapy (except that hormonal therapy for supportive care is permitted). Antiviral treatment is allowed, however interferon therapy must be stopped at least 4 weeks prior randomization.
  * Prior use of systemic investigational agents for HCC
  * Autologous bone marrow transplant or stem cell rescue within four months of start of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Overall survivals | 5 years

SECONDARY OUTCOMES:
Recurrence rates | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatobilliary Surgery, Affiliated Tumor of Guangxi University, Nanning, Guangxi, China